CLINICAL TRIAL: NCT06074497
Title: A Phase 1, First-in-Human, Multicenter, Open-Label, Dose Escalation Trial of KGX101 Monotherapy and in Combination with Envafolimab in Patients with Advanced or Metastatic Solid Tumors.
Brief Title: This is an Open Label, Two-part, Multicenter, Phase I Trial to Investigate the Safety, Tolerability, and PK of KGX101 Monotherapy and Combination Therapy with Envafolimab in Patients with Advanced or Metastatic Solid Tumors.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kangabio AUSTRALIA LTD PTY (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KGX101ST101
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- KGX101- Cohort -1 (Experimental): Dosage level: Dose level 1 Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort -1
- KGX101- Cohort 1 (Experimental): Dosage level: Dose level 2. Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort 1
- KGX101- Cohort 2 (Experimental): Dosage level: Dose level 3 Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort 2
- KGX101- Cohort 3 (Experimental): Dosage level: Dose level 4 Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort 3
- KGX101- Cohort 4 (Experimental): Dosage level: Dose level 5 Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort 4
- KGX101- Cohort 5 (Experimental): Dosage level: Dose level 6 Dose form: White-like lyophilized powder Route of administration: Intravenous
  Interventions: Drug: KGX101- Cohort 5
- KGX101 and Envafolimab (Active Comparator): Part B combination therapy KGX101 with Envafolibmab. Dose form: Injection Route to administration: Injection
  Interventions: Drug: KGX101 and Envafolimab

INTERVENTIONS:
Drug: KGX101- Cohort -1 — Single dose of 0.1, 0.3, 1μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort -1
Drug: KGX101- Cohort 1 — Single dose of 0.3, 1.0, 3.0μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort 1
Drug: KGX101- Cohort 2 — Single dose of 1, 1 and 3μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort 2
Drug: KGX101- Cohort 3 — Single dose of 1,3 and 6μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort 3
Drug: KGX101- Cohort 4 — Single dose of 1,3,12μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort 4
Drug: KGX101- Cohort 5 — Single dose of 2, 5 and 15 μg/kg of KGX101 every 3 weeks
  Arms: KGX101- Cohort 5
Drug: KGX101 and Envafolimab — Part B combination therapy KGX101 with Envafolibmab. 400mg to be injected subcutaneously with each target dose of KGX101 every 3 weeks. The dose escalation committee (DEC) may decide to increase the dosage to 600mg. based on PK, PD and safety data.
  Arms: KGX101 and Envafolimab

SUMMARY:
This is an open label, two-part, multicenter, multi-regional phase I trial to investigate the safety, tolerability, and PK of KGX101 monotherapy and combination therapy with Envafolimab in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study will enrol 54 participants depending on the number of dose escalations needed.

The study has 2 parts- Part A monotherapy dose escalation and Part B combination dose escalation. This study will assess KGX101 monotherapy (Part A) and in combination therapy with Envafolimab (Part B) by a standard 3+3 dose escalation design to identify the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D).

This study schedule will include a 28-day screening, a DLT observation period, followed by variable length study treatment period, 90-day safety follow-up after the last treatment, and survival follow-up every 90 days. Therefore, the total duration of participation will vary for each participant depending on total doses.

A priming dose is the initial lower dose(s) followed by escalation to the full treatment dose(s). Priming dose will be implemented in all cohorts. As the first 3 enrolled previously participants at 0.003 mg/kg didn't receive priming dose, the subsequent enrolled patients at this dose level will receive two priming doses before the target dose. Two priming doses of KGX101 with an dosing interval of 10 days will be recommended. Priming dose regimen may be adjusted by Dose Escalation Committee (DEC) based on the real-time safety, available PK and PD data.

The participants will receive KGX101 intravenous infusion at assigned escalating dose alone or in combined with 400mg Envafolimab every 3 weeks until disease progression or discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Any histologically or cytologically confirmed solid tumor malignancy that is locally advanced or metastatic and has failed standard therapy, or for which no further standard therapy exists.

   Part B- In addition to above for Part B, participants should be tumor PD-L1 expression negative or with PD-L1 expression too low to fit for the immune checkpoint inhibitor treatment or have had disease progression after immune checkpoint inhibitor treatment.
2. Age at least 18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1.
4. Has at least 1 measurable lesion per RECIST 1.1 (lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions).
5. Has adequate organ and bone marrow function as per the study (blood transfusion or use of use hematopoietic stimulating factor for correction within 14 days are not permitted):

   1. Hematologic: White blood cell (WBC) count ≥ 3 x 109/L; an absolute neutrophil count ≥ 1.5 x 109/L; a hemoglobin level > 90 g/L; and a platelet count ≥ 100 x 109/L;
   2. Adequate hepatic function as defined by:

      * Total bilirubin ≤ 1.5 times the ULN if no liver metastases or ≤ 2.5 times the ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases;
      * Aspartate transaminase (AST), alanine transaminase (ALT) and Alkaline phosphatase (ALP) levels ≤ 2.5 x the ULN or ≤ 5 x the ULN for patients with liver metastases;
      * Coagulation international normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x the ULN;
   3. Adequate renal function as defined by a serum creatinine ≤ 1.5 times the ULN concurrent with creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft-- Gault equation);
   4. Biochemistry: albumin ≥ 3.0g/dL
6. Willingness of men and women of reproductive potential to observe highly effective birth control for the duration of treatment and for 5 months following the last dose of study drug.
7. Paired pre-treatment archival tumor tissue within two years or fresh tumor biopsy and on-treatment fresh tumor biopsy will be optional. For participants of cutaneous malignant melanoma, paired pre-treatment archival tumor tissue and on-treatment fresh tumor biopsy should be mandatory
8. Life expectancy of approximately 3 months or longer in the opinion of the Investigator.
9. Provision of signed and dated written informed consent prior to any study-specific procedures, sampling, and analyses.

Exclusion Criteria:

1. Active known second malignancy with the exception of any of the following: adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer, breast cancer, papillary thyroid carcinoma; adequately treated stage I cancer from which the patient is currently in remission and has been in remission for ≥ 2 years; low risk prostate cancer with Gleason score < 7 and prostate-specific antigen <10ng/mL; any other cancer from which the patient has been disease-free survival for ≥ 5 years.
2. Patients with primary CNS malignancies.
3. A history of allogeneic tissue/solid organ transplant.
4. Any evidence of severe or uncontrolled systemic diseases, including:

   1. Active, uncontrolled systemic bacterial, viral, or fungal infection;
   2. uncontrolled hypertension (Systolic blood pressure more than equal to 160mHG or diastolic blod pressure more than equal to 100mm HG or poor compliance with anti-hypertensive agents;
   3. or active bleeding diatheses;
   4. Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]) or acute myocardial infarction within 6 months;
   5. Uncontrolled diabetes or poor compliance with hypoglycemic agents;
   6. The presence of chronically unhealed wound or ulcers;
   7. Other chronic diseases, which, in the opinion of the Investigator, could compromise safety of the patient or the integrity of study.
5. Active autoimmune disease requiring systemic treatment in the past 2 years.
6. Diagnosis of immunodeficiency, is on immunosuppressive therapy, or is receiving chronic systemic or enteric steroid therapy.
7. A history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
8. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
9. Active infection as determined by hepatitis B surface antigen and hepatitis B core antigen antibody, or hepatitis B virus DNA by quantitative polymerase chain reaction (qPCR) testing.
10. Active infection as determined by hepatitis C virus (HCV) antibody or HCV RNA by qPCR testing.
11. Major surgery (excluding placement of vascular access) within 4 weeks prior to the first dose of study drug.
12. Treatment with any of the following:

    1. Prior treatment with IL-12 therapy (any form, e.g. recombinant human, prodrug, intratumoral, etc.);
    2. Presence of CNS metastases that are symptomatic and/or require local CNS directed therapy (such as XRT or surgery) or increasing doses of corticosteroids within 2 weeks prior to the first dose of study drug. Except patients with treated brain metastases should be neurologically stable and receiving less than equal to 10mg per day of prednisone or equivalent prior to study entry;
    3. Investigational agent or anticancer therapy (including chemotherapy, biologic therapy, immunotherapy, anticancer Chinese medicine, or anticancer herbal remedy) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug;
    4. Radiotherapy within 2 weeks of the start of study treatment. A 1-week washout is permitted for palliative radiation (less than equal to two weeks of radiotherapy) to non-CNS disease;
    5. Received a live or live-attenuated vaccine within 30 days of the first dose of study drug; Note: Administration of killed vaccines or other formats are allowed;
    6. Diagnosis of immunodeficiency, on immunosuppressive therapy, or receiving chronic systemic or enteric steroid therapy (dose > 10 mg/day of prednisone or equivalent);
    7. Prior receipt of an allogeneic stem cell transplant or allogeneic CAR-T cell therapy;
13. Any unresolved toxicities from prior therapy greater than NCI CTCAE version 5.0 Grade 1 at the time of starting study drug with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy, and medical history conditions requiring maintenance therapy such as, but not limited to, hypothyroidism and adrenal insufficiency, where the principal investigator (PI) has the discretion to determine the appropriate severity classification at study screening, contingent upon the patient's screening labs not showing clinically significant abnormalities and meeting the eligibility requirements as per sponsor and site PI approval.
14. Electrocardiogram QT interval corrected for heart rate (QTc) > 470 msec, measured by Fridericia's formula [QTcF=QT/(RR0.33)]; or any of the following cardiac events within 6 months before screening: Myocardial infarction; unstable angina; unstable symptomatic ischemic heart disease; New York Heart Association class III or IV heart failure; Thromboembolic events (eg, pericardial effusion, restrictive cardiomyopathy, severe untreated valvular stenosis, or severe congenital heart disease).
15. Any illness, medical condition, organ system dysfunction, or social situation (including mental illness or substance abuse), that may interfere with a patient's ability to sign the ICF, adversely affect the patient's ability to cooperate and participate in the study, or compromise interpretation of study results.
16. Pregnant (confirmed by serum beta human chorionic gonadotropin [ HCG]) or lactating.
17. History of hypersensitivity to any of the study drug components; or history experienced grade ≥ 3 irAEs and leads to permanent discontinuation in prior immunotherapy.
18. Part B: participants who are not tolerant to immune checkpoint inhibitor therapy.
19. Participant is known or suspected of not being able to comply with the study protocol (e.g. because of alcoholism, drug dependency, or psychological disorder) or the participant has any condition for which, in the opinion of the Investigator, participation in the study would not be in the best interest of the participant (e.g. compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments. Or any other disease or clinically medical status that the investigator considers the patient is unstable or may affect their safety or study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment emergent Adverse events (TEAEs) | From baseline to 30 days after the last dose administration.
  TEAE will be collected to assess participants' safety after KGX101 treatment.
Number of participants with Dose Limiting Toxicities (DLTs) at week 4 | From Day 1 after the first dose of KGX101 full treatment to D21 post dose.
  DLT will be observed from start of treatment until 21 days post the first target dose treatment.
Number of participants with changes to clinical laboratory abnormalities | Screening to 90 days post last dose administration
  Any changes in values of the clinical chemistry, hematology, coagulation and urinalysis will be evaluated.
To estimate the Maximum tolerated dose of KGX101 monotherapy and combination therapy with Envafolimab. | From Day 1 after the first dose of KGX101 full treatment to D21 post dose.

SECONDARY OUTCOMES:
PK Parameters: Maximum Concentration (Cmax) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Time of maximum observed concentration (Tmax) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Area under the curve (AUC) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Half- life (T1 /2) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters- Trough concentration (Ctrough) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters- Systemic clearance (CL) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
Immunogenicity- Anti-drug antibody (ADA) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 hours after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Samples will be collected to assess the immunogeniccity after KGX101 treatment.
PK Parameters- Volume of distribution (Vd) | Part A- From pre-dose of the first dose of KGX101 full treatment to Day 90 hours after the first and 4th dose of full treatment; Part B- Predose and 72hrs (only 1st treatment)
  Part A- The PK schedule after the 1st and 4th injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Part B- PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
Number of participants with changes in the Investigator-assessed confirmed Best Overall Response (BOR) | From Day 1 after the first dose of KGX101 full treatment to D21 post dose.
Number of participants with changes in the Overall Response (ORR) | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.
Progression free survival (PFS) per RECIST 1.1 | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.
Overall survival | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.
Change in serum concentration of KGX101 and total IL-12 | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Jiang, Dr, Study Chair — Chief Executive Officer
Locations (3):
- Australia (3):
  - Pindara Private Hospital, Benowa, Queensland
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria

IPD SHARING:
Plan to Share IPD: No